CLINICAL TRIAL: NCT05010083
Title: The University of Michigan OWL (Online Wellness and Lifestyle) Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Nutrition Science Initiative (Other)
Responsible Party: Principal Investigator, Laura Saslow, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00192032
Record Dates: First submitted 2021-08-10; First posted 2021-08-18 (Actual); Last update posted 2022-10-24 (Actual); Status verified 2022-10

CONDITIONS: Obesity
Keywords: nutrition; Diet, Ketogenic; Diet, Carbohydrate-Restricted
MeSH Terms: conditions — Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- diet and lifestyle program (Experimental)
  Interventions: Behavioral: diet and lifestyle program

INTERVENTIONS:
Behavioral: diet and lifestyle program — See description of main arm.

SUMMARY:
The goal of this trial is to pilot test our existing very low carbohydrate diet intervention, adapted for young adults.

DETAILED DESCRIPTION:
Obesity increases the risk of a variety of illnesses such as heart disease, type 2 diabetes, cancer, sleep apnea, asthma, and depression. While advice from the Centers for Disease Control, American Heart Association, and the National Institutes of Health recommend a low-fat diet with a focus on whole grains and lean meats, research shows that a very low-carbohydrate diet may be more effective at reducing body mass index (BMI). Given the disconnect between recommendations and research, higher quality, long term, large trials are needed. In preparation for that research, the investigators plan to pilot test a very low-carbohydrate diet program, the OWL study (Online Wellness and Lifestyle Study), for 30 young adults followed over 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-25
* Obese (BMI ≥ 30)
* Sufficient control over diet
* Access to internet and texting
* Living in the United States
* Willing and able to follow intervention and complete measurements

Exclusion Criteria:

* Non-English speaking
* Pregnant, breastfeeding, or planning to be in the next 6 months
* Vegan or vegetarian
* Currently enrolled in weight loss program
* Taking medications known to cause weight loss or gain
* Taking glucose-lowering medications other than metformin
* Type 1 diabetes
* Cancer
* Heart failure
* Kidney failure
* History of eating disorders
* Untreated psychiatric disorder
* History of or planned weight loss surgery
* Consumption of greater than 30 alcoholic beverages per week

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2021-08-23 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Change in percent bodyweight | 4 months
  Measured with bodyweight scale

SECONDARY OUTCOMES:
Change in HbA1c | 4 months
  Measured with at-home finger prick analyzed in CLIA certified lab

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saslow LR, O'Brien A, Raymond K, Bayandorian H, Marriott D, Moskowitz JT, Daubenmier J, Bridges D, Cousineau CM, Griauzde DH. Feasibility and acceptability of an online multicomponent very low-carbohydrate intervention in young adult women with obesity: a pilot study. Pilot Feasibility Stud. 2024 Jul 29;10(1):102. doi: 10.1186/s40814-024-01525-0. PMID 39075617